CLINICAL TRIAL: NCT05533879
Title: The Effect of Yoga on Body Awareness and Kinesiophobia in Women With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61351342
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Women With Chronic Low Back Pain
Keywords: yoga, chronic low back pain, women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga group (Experimental): Women with having received a minimum of 17 points from the kinesiophobia questionnaire, have chronic low back pain and aged between 25-65
  Interventions: Other: Tele-yoga

INTERVENTIONS:
Other: Tele-yoga — Women with chronic low back pain will be taken to group-based Tele-Yoga sessions of 60 minutes three times a week for 4 weeks, in an internet-based telerehabilitation environment.

SUMMARY:
Chronic low back pain (CLBP) is the most common problem in the musculoskeletal system and causes disability. The prevalence of chronic low back pain is 80% in women. Although there are many causes of low back pain, it is often not possible to find the exact cause of the pain. The consequences of chronic low back pain include musculoskeletal problems, decreased sleep quality, decreased quality of life and limitation in activities of daily living, depression, anxiety, and decreased body awareness and kinesiophobia.

Kinesiophobia is defined as the fear of re-injury gained after injury, which reduces physical movement and activity. Patients with kinesiophobia develop the idea that movement will cause re-injury and add to pain. This situation leads to avoidance of physical activity and functional disability in the long term.

Body awareness, on the other hand, is the awareness of the messages that the brain receives from other parts of the body and from the outside. These messages that the person receives include not only his own body and movements, but also information such as the characteristics and locations of other objects in the environment. This information is blended over time and turns into experiences of the body.

Today, a rehabilitation method consisting of exercise programs, in which the active participation of the individual is ensured, is recommended, especially in the treatment approach to chronic low back pain. Within the scope of physiotherapy programs; heat applications and other physical therapy agents, exercise applications are recommended. Yoga is an alternative exercise practiced in CLBP as a body-mind exercise. Yoga is an easy-to-apply, non-invasive, cost-effective, scientifically proven practice.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a very important problem that affects many people in the world and has a negative impact on the economy. The prevalence of chronic low back pain is 80% in women and 70% in men. Although there are many causes of low back pain, it is often not possible to find the exact cause of the pain. Low back pain is classified as acute low back pain if it lasts for six weeks, subacute low back pain between six weeks and three months, and chronic low back pain if it lasts for more than three months.

CLBP is a complex problem that persists for a long time without a cause and is the most common in the musculoskeletal system and causes disability. Although low back pain is seen more frequently in women, its distribution varies according to gender when different etiologies are examined. Among the consequences of chronic low back pain are depression, anxiety, anxiety disorder, loss of muscle flexibility and power losses, joint disc degenerations, circulation problems, musculoskeletal system problems, decrease in sleep quality, decrease in quality of life and limitation in daily living activities, along with the pain-spasm cycle. decreased body awareness and kinesiophobia.

Kinesiophobia is defined as an excessive fear of re-injury that can be gained after a painful injury and reduces physical movement and activity. Patients with kinesiophobia develop the idea that movement will cause re-injury and add to pain. This leads to avoidance of physical activity in the long term, functional disability, depression and a decrease in quality of life.

Body awareness is a special form of consciousness. In neuroscience, body awareness is the brain's awareness of messages it receives from other parts of the body and from the outside. These messages that the person receives include not only his own body and movements, but also information such as the characteristics and locations of other objects in the environment. This information is blended over time and turns into experiences of the body.

Today, a rehabilitation method consisting of intense exercise programs, in which the active participation of the individual is ensured, is recommended instead of the passive treatment method, especially in the treatment approach to the individual with chronic low back pain. Early mobilization and exercise have been found to be beneficial in individuals with low back pain. Different physiotherapy programs are recommended for individuals with CLBP. Within the scope of physiotherapy programs; heat applications and other physical therapy agents, exercise applications are recommended. Exercise applications are especially recommended for low back pain.

Yoga is an alternative exercise applied in CLBP as a body-mind exercise. It has been reported that yoga has been used frequently in recent years because it provides core-stabilization, increases flexibility and balance, and controls pain with relaxation exercises.

Yoga is an easy-to-apply, non-invasive, low-cost, scientifically proven practice, and with the holistic well-being it brings, it promises hope for both physical and mental illnesses. When the literature is examined, there are studies that include the effects of yoga on quality of life, sleep quality, pain intensity, functional status, balance in people with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Having received a minimum of 17 points from the kinesiophobia questionnaire
* Being between the ages of 25 and 65 and being a woman
* Having a complaint of low back pain for at least 6 months
* Not having cognitive, cognitive and mental problems

Exclusion Criteria:

* Having had surgery involving the spine.
* Being involved in any yoga group for the last 6 months
* Actively exercising regularly
* A previous or existing neurological disorder

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with chronic low back pain
Enrollment: 50 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | 10 minutes
  This form was prepared by the researchers to obtain the demographic data of the people participating in the study. In this form, information about the age, gender and occupation of the participants is recorded.
Visual Analog Scale (VAS) | 2 minutes
  When Visual Analog Scale (VAS) is used, I have no pain at one end, very severe pain is written on the other end, and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.
Body Awareness Questionnaire | 20 minutes
  The questionnaire is based on people's ratings of the situations they feel about themselves. After reading each statement, the number 1 to 7 is marked in the space to the left of the statement, which is appropriate for the person who filled out the questionnaire. The most accurate answer is the experience of the person filling out the questionnaire.
Tampa Kinesiophobia Scale | 20 minutes
  It is a 17-item scale developed to measure fear of movement/re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. As a result of the survey, the person gets a total score between 17-68 according to the answers he/she gives. The higher the score the person gets on the scale, the higher the kinesiophobia.
  shows that.

CONTACTS AND LOCATIONS:
Overall Officials: tuba kolaylı, MSc., Study Director — Uskudar University; Aleyna Yaren Bayrak, B.S., Principal Investigator — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided